CLINICAL TRIAL: NCT01357590
Title: Evaluation of the Vascutek Ltd. Thoracic Endovascular Stent Graft System (ThoraflexTM)in the Treatment of Aneurysm or Penetrating Ulcer of the Descending Thoracic Aorta
Brief Title: Evaluation of Thoraflex in the Treatment of Aneurysm or Penetrating Ulcer of the Descending Thoracic Aorta
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAA-001
Record Dates: First submitted 2011-05-17; First posted 2011-05-20 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Aortic Aneurysm, Thoracic; Penetrating Aortic Ulcers (PAUs)
Keywords: aneurysm, penetrating ulcer, descending thoracic aorta
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Penetrating Atherosclerotic Ulcer; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Thoracic Endovascular Stent Graft System (ThoraflexTM) — Thoracic Endovascular Stent Graft System

SUMMARY:
ThoraflexTM is designed for the treatment of aneurysm or penetrating ulcer of the descending thoracic aorta. Each system is advanced from a transfemoral or transiliac approach over a 0.035" guidewire and positioned under fluoroscopic control. If necessary, an arterial conduit technique may be required to allow access to the arterial system. The soft tapered tip allows atraumatic insertion into the vessel, while the catheter and sheath are designed to provide excellent flexibility and control through tortuous arterial anatomy.

Each individual stent graft device is supplied sterile and pre-loaded in a single-use delivery system. The stent graft is a self-expanding endoprosthesis constructed of a thin wall woven polyester and nitinol ring stents, which are attached to the fabric with braided polyester sutures. The delivery system central catheter is a stainless steel braided co-extrusion of polytetrafluoroethylene (PTFE) and polyester elastomer, designed to provide significant torque control and strength, while also maintaining superior flexibility. The outer sheath is made in a tri-layer construction consisting of a PTFE liner, a stainless steel flat braid layer and a polyester elastomer outer jacket with a hydrophilic lubricant coating. These materials provide very low friction force during device insertion and deployment together with enhanced flexibility of the delivery system. The handle components are moulded from thermoplastic polyurethane.

The materials of the endoprosthesis are identical to those of the current Conformité Européenne (CE) marked Vascutek Ltd. AnacondaTM Stent Graft System intended for abdominal aortic aneurysm repair. The materials of the delivery system are well established in medical applications. The design of ThoraflexTM is based on the same principles as other clinically established thoracic endovascular devices. The endoprosthesis is constructed of self-expanding nitinol stents and a polyester tube graft. Four proximal hooks anchor the endoprosthesis within the aorta. Unlike existing thoracic endovascular devices, the delivery system of ThoraflexTM allows repositioning of the endoprosthesis so that the optimal deployment position can be enhanced.

The intended use of ThoraflexTM is the treatment of aneurysm or penetrating ulcer of the descending thoracic aorta, which is identical to other CE approved thoracic endovascular devices.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged > 18 years
2. Subject has a life expectancy of at least 12 months
3. The Subject must meet at least one of the following:

   1. Descending thoracic fusiform aneurysm, 50mm in diameter or greater. ONLY FOR FRENCH SITES: Descending thoracic fusiform aneurysm, 5.5cm in diameter or greater.
   2. Descending thoracic aneurysm that is 4cm or more in diameter that has increased in size by 0.5cm in last 6 months. ONLY FOR FRENCH SITES: Descending thoracic aneurysm that is 4cm or more in diameter that has increased in size by 1cm in the last year
   3. Descending thoracic aneurysm with a maximum diameter that exceeds two times the diameter of the non-aneurysmal, adjacent aorta
   4. Saccular aneurysm in the descending thoracic aorta or Penetrating Atherosclerotic Ulcers (PAUs). ONLY FOR FRENCH SITES: Saccular aneurysm in the descending thoracic aorta, Penetrating Atherosclerotic Ulcers (PAUs) with associated Intramural Haematoma, or Atherosclerotic Giant PAU
4. Subject must have proximal and distal aortic neck suitable for stent graft placement with vessel diameter ranging between 22.0 - 35.0 mm.
5. The length of attachment zones will depend on the intended stent graft diameter. For left subclavian artery (LSA) in superior position: The proximal attachment zone should be 10mm for 28mm graft, 11mm for 30mm, 12mm for 32mm - 34mm grafts, 14mm for 36mm - 38mm grafts and 15mm for 40mm graft. For LSA in non-superior position: The proximal attachment zone should be 15mm for 28mm graft, 17mm for 30mm, 20mm for 32mm - 34mm grafts, 23mm for 36mm - 38mm grafts and 25mm for 40mm graft. The distal attachment zone should be 40mm.
6. The diagnosis is confirmed as thoracic aortic aneurysm or PAU by contrast enhanced CT obtained within the three months prior to implant.
7. Access vessels: Adequate iliac/femoral access -able to accommodate 23 (7.7 mm) or 25 OD French size (8.3 mm) introducer systems, with or without the use of an arterial conduit.
8. Subject is able and willing to comply with the protocol and associated follow-up requirements
9. Subject or legal representative must have agreed to participate voluntarily and have signed and dated an Ethics Committee/Ethical Review Board approved Patient Informed Consent form.

Exclusion Criteria:

1. Subject has any of the following conditions in his/her descending thoracic aorta:

   1. Dissections - acute or chronic, in ascending or descending aorta
   2. Acute Transection or Acute Traumatic Injury
   3. Pseudoaneurysm (false aneurysm)
   4. Symptomatic Aneurysm, including ruptured lesions
2. Subject's proximal neck diameter measures < 22.0 or > 35.0 mm.
3. Subject's distal neck diameter measures < 22.0 or > 35.0 mm.
4. Subject has prohibitive calcification (>50% circumferential calcification), occlusive disease, or tortuosity of intended fixation sites.
5. Subject has circumferential thrombus (>50%) in region of intended fixation sites.
6. Subject has an increasing tapered proximal neck with ≥3mm increase in diameter from proximal fixation site to the aneurysm.
7. Subject has a decreasing tapered distal neck with ≥3 mm increase in diameter from distal fixation site to the aneurysm.
8. Subject's aneurysm or distal thoracic aortic neck angle precludes advancement of the introduction system and device.
9. Subject has an anatomical variance which would compromise circulation to the carotids, vertebral, or innominate arteries after device placement that is not amenable to subclavian revascularisation. This would not apply to Subjects with occluded celiac arteries.
10. Subject is pregnant.
11. Subject is morbidly obese preventing adequate x-ray visualization of the aorta.
12. Subject has known or suspected connective tissue disorder (e.g., Marfan's syndrome, Ehlers-Danlos syndrome).
13. Subject has a blood coagulation disorder or bleeding diathesis in which the treatment cannot be suspended for one week pre and post repair.
14. Subject has coronary artery disease with unstable angina and who has not received coronary revascularisation within the last 3 months.
15. Subject has chronic obstructive pulmonary disease requiring the routine need for oxygen therapy outside the hospital setting (e.g., daily or nightly home use).
16. Subject is in acute renal failure or renal insufficiency with a creatinine ≥ 2.5 mg/dL and is not on renal replacement therapy or dialysis.
17. Subject has active systemic infection and/or mycotic aneurysms.
18. Subject has had a stroke within 3 months of the treatment date.
19. Subject has less than one-year life expectancy as evidenced by factors prohibiting major medical intervention (e.g., presence of malignant tumour, advanced age, etc.).
20. Subject is participating in another research study.
21. Subject has a co-existing abdominal aortic aneurysm (AAA) in which the investigator believes requires concomitant treatment within 45 days.
22. Subject has had a prior AAA repair (endovascular or surgical) that was performed less than 6 months prior to enrolment.
23. Subject has had a prior endovascular repair (e.g., stent, stent-graft) in the descending thoracic aorta. The device may not be placed within any prior surgical graft.
24. Subject has an untreatable allergy or sensitivity to contrast media or device components.
25. Subject has been admitted to the hospital for a major surgical or medical procedure within45 days of the planned procedure or is planning to undergo other major surgical or medical procedure within 45 days post implantation (e.g., coronary artery bypass graft [CABG], organ transplantation, etc.). This excludes any planned procedures for the prospective stent-graft placement (e.g. common carotid to left subclavian transposition/bypass, left carotid to axillary bypass, etc. are acceptable. Carotid-carotid bypasses are not permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Successful aneurysm/PAU treatment, defined as a composite endpoint of Subjects who have successful delivery and deployment of the ThoraflexTM at the initial procedure and are free from the following; | (less than or equal to) 365 days post-procedure
  1. Aneurysm growth (greater than or equal to) 5mm from baseline measurement
  2. Post-operative interventions to correct type I or III endoleaks
  3. Conversion to open surgical repair
  4. Failed patency of the stent graft
  5. Migration requiring secondary intervention
  6. Significant failure of stent graft integrity
  7. Aneurysm rupture

SECONDARY OUTCOMES:
Incidence of type I or III endoleak. The incidence of Subjects with freedom from type I and III endoleaks will be the focus of assessments; however type II and IV endoleaks will be recorded and evaluated for rates of occurrence | First 24 hour post-operative period (defined on procedural angiography)
Stent graft patency, described as the presence of blood flow within the graft as determined through imaging analysis | First 24 hour post-operative period (defined on procedural angiography)
Conversion to surgical repair | First 24 hour post-operative period (defined on procedural angiography)

CONTACTS AND LOCATIONS:
Locations (28):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc (UCL), Brussels
  - UZ Gent, Ghent
  - UZ (Universitair Ziekenhuis) Leuven, Leuven
- Canada (4):
  - Peter Lougheed Centre, Calgary
  - Institute University de Cardiologie et de, Québec
  - Sunnybrook Health Sciences Centre, Toronto
  - St Michael's Hospital, Toronto
- France (3):
  - Service de Chirurgie Cardaque et Vasculaire, Bordeaux
  - Hopital Europeen Georges Pompidou, Paris
  - Service de Radiologie, Toulouse
- Germany (6):
  - RWTH Aachen, University Hospital Aachen, Aachen
  - Harzzentru der Universitatsklinik Koln, Cologne
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Department of Vascular Medicine, Hamburg
  - MH Hannover, Hanover
  - Klinikum rechts der Isar, Munich
- Italy (3):
  - Universita di Bologna, Bologna
  - University of Florence, Florence
  - Dipartimento Cardioscienze, Rome
- Netherlands (5):
  - VUmc, Department of Surgery, Amsterdam
  - Academic Medical Centre (AMC), Department of Surgery, Amsterdam
  - Medisch Specturm Twente, Department of Surgery, Enschede
  - University of Maastricht, Department of Surgery, Maastricht
  - Erasmus Medical Centre, Department of Surgery, Rotterdam
- United Kingdom (4):
  - Leeds General Infirmary, Leeds, England
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Western Infirmary, Glasgow
  - St Thomas' Hospital, London